CLINICAL TRIAL: NCT05000138
Title: FDG Digital PET/CT as First Line Investigation for Giant Cell Arteritis
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Gad Abikhzer, Associate Professor, Jewish General Hospital
Other Study IDs: MP-05-2021-2846
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Giant Cell Arteritis; Vasculitis
Keywords: FDG PET/CT; digital PET
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: FDG PET/CT — Patients with suspected giant cell arteritis, of which FDG PET/CT is indicated for diagnosis of large vessel involvement, will have the small cranial arteries analyzed for involvement.

SUMMARY:
Giant cell arteritis (GCA) causes inflammation of the arteries and can lead to serious complications such as blindness, necessitating rapid diagnosis and treatment. Although older technology non-digital PET/CT scans are routinely used for the diagnosis of GCA in large arteries, they have not been able to reliably detect inflammation of the small arteries responsible for blindness. Recent technological advances have enabled PET/CT imaging of millimetric disease in the body, which are now able to resolve small arteries. In the proposed research study, patients who are suspected by their doctors to have GCA will undergo an ultrasound of the temporal arteries, and digital PET/CT scan after injection of radioactive glucose. Digital PET/CT scans will be interpreted for the presence of abnormal uptake in the large and small arteries, as well as for the presence of other causes of the patient's symptoms. The diagnostic accuracy of PET/CT and ultrasound will be evaluated with respect to an expert panel diagnosis of giant cell arteritis and compared. Results will be adjusted for lack of a perfect reference test using advanced statistics. The goal will be to see if digital PET/CT can become a single, integrated test to diagnose this disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years, capable and willing to provide informed consent and can tolerate PET/CT.
* ESR ≥ 50 mm/h and/or CRP ≥ 10mg/L within 1 week of PET/CT referral.
* New suspected giant cell arteritis according to at least one of the following criteria:

Cranial GCA symptoms (new-onset localized headache, scalp or temporal artery tenderness, ischemia-related vision loss, masseter pain on prolonged mastication) PMR symptoms: shoulder and/or hip girdle pain associated with inflammatory stiffness.

Suspected large-vessel vasculitis based on angiography, MRA, or CTA.

Exclusion Criteria:

* Initiation of corticosteroid or immunosuppressive therapy >4 days before PET/CT.
* Prior TAB or treated GCA with suspected relapse.
* Non-fasting or hyperglycemia (>11.1 mmol/L) resulting in altered FDG biodistribution.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected GCA
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance | 2 years
  of Digital PET/CT and DUS for the diagnosis of GCA

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (3):
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHUS, Sherbrooke, Quebec
- Université Bourgogne Europe, Centre Georges-François Leclerc, Dijon, France
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No